CLINICAL TRIAL: NCT01488955
Title: Immediate vs. Conditional Use of Antibiotics in Uncomplicated Urinary Tract Infection (UTI) - a Comparative Effectiveness Study in General Practice (ICUTI)
Brief Title: Immediate vs. Conditional Use of Antibiotics in Uncomplicated Urinary Tract Infection (UTI) - ICUTI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut fuer anwendungsorientierte Forschung und klinische Studien GmbH (Other)
Collaborators: University Medical Center Goettingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20110512-BG
Record Dates: First submitted 2011-12-07; First posted 2011-12-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Urinary Tract Infection
Keywords: bacterial infection
MeSH Terms: conditions — Urinary Tract Infections; Bacterial Infections | interventions — Ibuprofen; Fosfomycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibuprofen (Experimental): Ibuprofen 400 mg oral once daily from day 0 for 3 days, placebo granulate oral day 0
  Interventions: Drug: Ibuprofen
- Fosfomycin-Trometamol (Experimental): Fosfomycin-Trometamol (Monuril) 3 g granulate oral at day 0, placebo to Ibuprofen once a day from day 0 for 3 days
  Interventions: Drug: Fosfomycin-Trometamol

INTERVENTIONS:
Drug: Ibuprofen — 400 mg oral once a day from day 0 for 3 days
  Arms: Ibuprofen
Drug: Fosfomycin-Trometamol — 8 g granulate with 3 g Fosfomycin-Trometamol oral once at day 0, placebo to Ibuprofen once a day oral from day 0 for 3 days
  Other Names: Monuril
  Arms: Fosfomycin-Trometamol

SUMMARY:
In this study, patients with uncomplicated urinary infection are investigated. It is investigated if treatment of only symptoms of the uncomplicated urinary infection is as effective as treatment with antibiotics with respect to the outcome of the urinary infection. If this is the case, the use of antibiotics in the treatment of uncomplicated urinary infections might be reduced.

Secondary aim of the study is the safety evaluation of both treatment strategies with respect to SAEs during treatment. Additionally, relapse frequency after 28 days is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Women (18 - 65 years)
* Symptoms of uncomplicated urinary tract infection: dysuria, frequency/urgency of micturition, and/or low abdominal pain
* written informed consent

Exclusion Criteria:

* fever (> 38,0)
* pain on renal bed percussion
* signs of complicated urinary tract infection
* urinary tract infection within the last two weeks
* antibiotic intake within the last 7 days
* repeated intake of pain medication (i.e. ibuprofen, diclofenac) within the last 24 hours, or continuous pain medication
* known pregnancy/lactation period
* current immunosuppressive therapy
* known renal insufficiency
* known renal abnormalities
* current urine catheterization
* serious neurological diseases
* limited condition due to other disorders
* contraindications towards trial medication
* current/anamnestic gastrointestinal haemorrhagia
* known allergy towards trial medication
* current intake of drugs potentially interacting with trial medication (i.e. oral corticosteroids, anticoagulates)
* poor communication/cooperation skills
* disability to understand trial information, poor German language skills
* current participation in another clinical trial or clinical trial participation within the last 4 weeks

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
number of additional treatments with antibiotics combined with number of symptoms | day 0-28
  The study outcome is considered as positive, if the interventional group where only symptoms were treated has less additional treatments with antibiotics as the interventional group, where antibiotics are given from day 0 on. Additionally, the interventional group where only symptoms were treated has to be non inferior with respect to number of symptoms.

SECONDARY OUTCOMES:
number of defined daily doses of antibiotics | day 0-28
number of SAEs | day 0-28
number of relapses | day 0-28
number of patients without symptoms | day 4 and day 7
symptom load (AUC) | day 0-4
symptom load | day 0-7
symptoms load with regard to specific symptoms | day 0-7
activity impairment assessment | day 0-7

CONTACTS AND LOCATIONS:
Overall Officials: Eva Hummers-Pradier, Prof., Principal Investigator — Abt. Allgemeinmedizin, Universitätsmedizin Göttingen, Humboldtallee 38, 37073 Göttingen
Locations (2):
- Germany (2):
  - Univercity Medical Center Goettingen, Göttingen
  - MHH Hannover, Hanover

REFERENCES:
- [Derived] Sachdeva A, Rai BP, Veeratterapillay R, Harding C, Nambiar A. Non-steroidal anti-inflammatory drugs for treating symptomatic uncomplicated urinary tract infections in non-pregnant adult women. Cochrane Database Syst Rev. 2024 Dec 19;12(12):CD014762. doi: 10.1002/14651858.CD014762.pub2. PMID 39698942
- [Derived] Gagyor I, Bleidorn J, Kochen MM, Schmiemann G, Wegscheider K, Hummers-Pradier E. Ibuprofen versus fosfomycin for uncomplicated urinary tract infection in women: randomised controlled trial. BMJ. 2015 Dec 23;351:h6544. doi: 10.1136/bmj.h6544. PMID 26698878
- [Derived] Gagyor I, Hummers-Pradier E, Kochen MM, Schmiemann G, Wegscheider K, Bleidorn J. Immediate versus conditional treatment of uncomplicated urinary tract infection - a randomized-controlled comparative effectiveness study in general practices. BMC Infect Dis. 2012 Jun 28;12:146. doi: 10.1186/1471-2334-12-146. PMID 22742538